CLINICAL TRIAL: NCT00600288
Title: A Multi-Center, Parallel-Group, Double-Masked, Randomized, Placebo-Controlled Study of the Effects of Diquafosol Tetrasodium Ophthalmic Solution, 2% and Placebo in Subjects With Dry Eye Disease
Brief Title: Study of the Effect of Diquafosol Tetrasodium Ophthalmic Solution, 2% Versus Placebo in Dry Eye Subjects (P08634)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P08634; 03-111
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2014-12

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: diquafosol tetrasodium Ophthalmic Solution, 2%
- 2 (Placebo Comparator)
  Interventions: Drug: Non-preserved saline solution (Placebo)

INTERVENTIONS:
Drug: diquafosol tetrasodium Ophthalmic Solution, 2% — 1-2 drops administered in each eye 4 times a day for 6 weeks
  Arms: 1
Drug: Non-preserved saline solution (Placebo) — 1-2 drops administered in each eye 4 times a day for 6 weeks
  Arms: 2

SUMMARY:
The purpose of this pilot study is to evaluate the effect of diquafosol tetrasodium Ophthalmic Solution, 2% in dry eye subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to any study procedures being performed.
* Have a best corrected visual acuity (BCVAof +0.7 or better.
* Have a history of dry eye (keratoconjunctivitis sicca) in both eyes
* Have ongoing dry eye disease, in the same qualifying eye or both eyes.

Exclusion Criteria:

* Have previously had LASIK refractive surgery.
* Use of topical ophthalmic medications, preps, gels and lid scrubs during study.
* Have had penetrating intraocular surgery in the past 90 days.
* Have had other ocular surface surgery (e.g., refractive, pterygium) within the past year.
* Have a diagnosis of an on-going ocular infection, clinically significant blepharitis, lid margin inflammation, Stevens-Johnson syndrome or pemphigoid.
* Any serious ocular systemic disease or uncontrolled medical condition.
* Exposure to any investigational drug within 30 days of study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change in fluorescein staining scores of the cornea | 6 weeks

SECONDARY OUTCOMES:
Safety and Tolerability | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Saiid Davari, Study Director — Merck Sharp & Dohme LLC